CLINICAL TRIAL: NCT06993246
Title: Does Supplemental Contrast-enhanced Mammography Have a Benefit in Women With a Personal History of Breast Cancer and Dense Breast Tissue? A Prospective Cohort Study.
Brief Title: Contrast-enhanced Mammography in Women With a Personal History of Breast Cancer and Dense Breast Tissue: Benefit?
Acronym: CEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jean Seely (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor-Investigator, Jean Seely, Physician Medical Imaging, Ottawa Hospital Research Institute
Organization: Ottawa Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OHSN- REB 20240828-01H
Record Dates: First submitted 2025-05-14; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Mammography screening; Contrast-Enhanced Mammography; Dense breasts
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study follows a **prospective cohort design**, where eligible participants are recruited and followed over time to evaluate the outcomes of Contrast-Enhanced Mammography (CEM) in comparison to traditional screening methods like ultrasound and MRI. Participants are women aged 50-69 years with dense breast tissue and a personal history of breast cancer. They will undergo CEM as part of their routine screening process. The study aims to assess key outcomes, including cancer detection rates, biopsy results, patient acceptance, and screening wait times. Data will be collected on screening outcomes, including abnormal interpretation rates, positive predictive values, and follow-up results over two years. The study also compares the performance of CEM with historical data from previous screening modalities.
Masking Description: There are no additional parties masked in this clinical trial. The study is open-label, meaning that participants, care providers, investigators, and outcomes assessors are all aware of the intervention being performed (Contrast-Enhanced Mammography). No masking of roles is applied in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- **Contrast-Enhanced Mammography for Supplemental Breast Cancer Screening** (Experimental): This arm involves participants undergoing Contrast-Enhanced Mammography (CEM) as a supplemental screening method for breast cancer. CEM combines standard mammography with iodinated contrast medium to improve lesion visualization and tumor detection, particularly in women with dense breast tissue. Participants will receive CEM during a single visit at the Rose Ages Breast Health Centre, and their results will be evaluated for cancer detection, abnormal interpretation rates, and biopsy outcomes.
  Interventions: Diagnostic Test: Contrast-Enhanced Mammography (CEM)

INTERVENTIONS:
Diagnostic Test: Contrast-Enhanced Mammography (CEM) — The intervention involves the use of contrast-enhanced mammography (CEM) to supplement standard mammography for breast cancer screening. This method utilizes iodinated contrast medium to enhance the visualization of breast lesions by assessing tumor neovascularization. CEM will be offered to women with dense breast tissue who are currently awaiting supplemental ultrasound screening. It is designed to be performed in conjunction with regular mammography, offering a more efficient and cost-effective alternative to MRI, with comparable sensitivity in detecting breast cancer. Participants will undergo the CEM procedure in a single visit, allowing for reduced wait times and improved detection rates compared to traditional methods. The procedure is well-tolerated, with minimal side effects, and provides a quicker and more accessible option for supplemental breast cancer screening.

SUMMARY:
This study aims to assess the effectiveness of Contrast-Enhanced Mammography (CEM)as an alternative to traditional ultrasound for breast cancer screening in women with dense breasts and a personal history of breast cancer. CEM combines standard mammography with a contrast agent to better detect tumors, particularly in women with dense tissue where traditional mammograms may miss signs of cancer. The study will compare CEM with ultrasound and MRI to determine its accuracy in detecting cancer, reduce wait times for screening, and provide a more affordable option than MRI. Women who participate will have their screening done in one visit, improving convenience and access. The study will track cancer detection rates, biopsy results, and patient satisfaction over two years to evaluate the benefits of CEM for early breast cancer detection.

DETAILED DESCRIPTION:
Primary Outcome Measure: 1. Detection Rate of Breast Cancer The primary outcome measure is the detection rate of breast cancer in women with dense breast tissue using contrast-enhanced mammography (CEM). The sensitivity, specificity, and overall accuracy of CEM in detecting malignancies will be compared to conventional mammography and ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting at Rose Ages Breast Health Center, who are currently waiting for supplemental screening Ultrasound, according to pre-established guidelines at TOH for supplemental screening.
* Women ages 50-69 years of age
* Those willing to participate in the study, sign an informed consent and undergo IV iodinated contrast injection
* Women with dense breasts (category C or D) and normal mammograms (BI-RADS 1 or 2)
* No evidence of renal disease

Exclusion Criteria:

* Patients with renal insufficiency (reduced eGFR <20ml/min)
* Previous allergic reactions to Iodine-based contrast.
* Prior contrast allergy (CT contrast)
* Thyroid Disease

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — * Women presenting at Rose Ages Breast Health Center, who are currently waiting for supplemental screening Ultrasound, according to pre-established guidelines at TOH for supplemental screening.
  * Women ages 50-69 years of age
  * Those willing to participate in the study, sign an informed consent and undergo IV iodinated contrast injection
  * Women with dense breasts (category C or D) and normal mammograms (BI-RADS 1 or 2)
  * No evidence of renal disease
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Detection Rate of Breast Cancer | Three years from the study start date.
  The primary outcome measure is the detection rate of breast cancer in women with dense breast tissue using contrast-enhanced mammography (CEM). The sensitivity, specificity, and overall accuracy of CEM in detecting malignancies will be compared to conventional mammography and ultrasound.

SECONDARY OUTCOMES:
Lesion Characterization | Up to one year.
  Assessment of the ability of CEM to accurately characterize breast lesions in terms of malignancy (benign or malignant). This will be evaluated by comparing CEM findings with biopsy results.
Patient Experience | Immediate post-procedure.
  A patient-reported survey measuring comfort, satisfaction, and perceived usefulness of CEM compared to traditional mammography.

OTHER OUTCOMES:
Procedure Safety | Three years from the study start date.
  Monitor and report any adverse events, including allergic reactions to the contrast medium and other side effects during and after the procedure.
Cost-Effectiveness | Three years from study start.
  Evaluation of the cost-effectiveness of CEM compared to conventional breast cancer screening methods, taking into account the costs of imaging, diagnosis, and follow-up procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jean Seely Principal Investigator,, MD FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared.